CLINICAL TRIAL: NCT05472831
Title: Optimizing Cognition Via Exercise and Nutrition
Acronym: OCEAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: University of Illinois at Chicago (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 5P30AG022849-18 (NIH); 5P30AG022849-18 (NIH)
Record Dates: First submitted 2021-12-17; First posted 2022-07-25 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Cognitive Function 1, Social
Keywords: Physical activity; Diet; Health disparities
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BAILAMOS dance program plus MIND diet (Experimental): BAILAMOS dance program plus MIND diet: Includes a 6-month, twice a week x 60 minutes/session, virtually delivered Latin dance program plus a 60 minute MIND diet session per week.
  Interventions: Behavioral: BAILAMOS dance program plus MIND diet
- BAILAMOS dance program plus Health Education (Experimental): BAILAMOS dance program plus Health Education: Includes a 6-month, twice a week x 60 minutes/session, virtually delivered Latin dance program plus a 60 minute health education session per week.
  Interventions: Behavioral: BAILAMOS dance program plus Health Education

INTERVENTIONS:
Behavioral: BAILAMOS dance program plus MIND diet — The refined BAILAMOS program is a Latin dance, Spanish-language intervention that encompasses six dance styles (Merengue, Cha Cha Cha, Bachata, Salsa, Cumbia and Samba). The program meets twice weekly for 60 minutes per session during 6-months via Zoom. The experimental group will also receive one, 60 minute MIND diet session per week.
  Arms: BAILAMOS dance program plus MIND diet
Behavioral: BAILAMOS dance program plus Health Education — The refined BAILAMOS program is a Latin dance, Spanish-language intervention that encompasses six dance styles (Merengue, Cha Cha Cha, Bachata, Salsa, Cumbia and Samba). The program meets twice weekly for 60 minutes per session during 6-months via Zoom. The experimental group will also receive one, 60 minute Health Education session per week.
  Arms: BAILAMOS dance program plus Health Education

SUMMARY:
Investigators propose to test the preliminary efficacy of the refined BAILAMOS™ Latin dance program plus a culturally tailored MIND diet (Mediterranean-DASH diet intervention for neurodegenerative delay) program on cognitive function among older Latinos (ages 50+) at risk of cognitive decline. This project will test whether participants randomized to the BAILAMOS™ Latin dance plus MIND diet experience better cognitive outcomes than participants randomized to the BAILAMOS™ Latin dance plus a health education program.

DETAILED DESCRIPTION:
By 2060, the prevalence of Alzheimer's disease (AD) in Latinos is projected to increase by 832%. There is an urgent need to create non-pharmacological interventions to reduce the risk of AD among Latinos. Physical activity (PA) and diet interventions (e.g. Mediterranean-DASH Intervention for Neurodegenerative Delay (MIND)) have been shown to decrease the incidence of AD. Behavioral interventions that concomitantly target physical activity (PA) and diet have shown an improvement in cognitive function; however, these studies have not been conducted in older Latinos nor have they included culturally appropriate interventions. The need to test culturally appropriate PA and diet interventions that have the potential to reduce the loss of cognitive function in older Latinos, a group at elevated risk of health disparities, is of high public health importance. OCEAN (Optimizing Cognition via Exercise and Nutrition) is a 6-month multidomain (Latin dance plus MIND DIET) intervention delivered virtually to middle-aged and older Latinos. The investigators propose a pilot randomized controlled trial to test the preliminary efficacy of the refined BAILAMOS™ Latin dance program plus MIND (Mediterranean-DASH diet intervention for neurodegenerative delay)- a new program tailored for the protection of the brain. The impact of the combined program (intervention group (IG)) will be compared to a BAILAMOS™ plus health education (control group (CG)) on cognitive performance among middle-aged to older Latinos at risk of cognitive decline.

ELIGIBILITY:
Inclusion Criteria:

1. age 50 years and older
2. self-identification as Latino/Hispanic
3. ability to understand Spanish
4. score of >21 on the Telephone Interview of Cognitive Status (TICs-m)
5. <3 days or <90 minutes of moderate-to-vigorous physical activity per week
6. self-report having a cardiovascular disease (CVD) OR at least one CVD risk factor (i.e., hypertension, hyperlipidemia, diabetes, obesity, current smoker, or family history of CVD) OR family history of Alzheimer's disease
7. administer EASY questionnaire-yes to any question means they will need medical clearance)
8. Suboptimal diet assessment <8
9. must be able to attend a one-hour orientation before the start of the intervention
10. have access to a tablet or computer with internet access.

Exclusion Criteria:

1. significant physical illness or medical condition that would preclude participation in a dance program
2. current or past history of a significant psychiatric condition that would interfere with participation in the study
3. presence of self-reported uncontrolled cardiovascular disease or uncontrolled diabetes mellitus
4. severe chronic obstructive pulmonary disease
5. recent healing or unhealed fracture(s)
6. had recurrent falls in the past 12 months
7. hip or knee replacement
8. participated in a structured dance program for 2 or more days in the past month
9. Sub-optimal diet assessment >8
10. Cannot attend a one-hour orientation before the start of the intervention
11. Travel for more than 2-weeks throughout course of intervention and do not have access to internet

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2024-10-19 (Actual); Study Completion 2024-10-19 (Actual)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) | Change in scores from baseline to post-intervention 6 months
  MoCA version 8.1 Blind will be used to assess global cognition. The MoCA-BLIND assesses different cognitive domains such as attention and concentration, memory, language, conceptual thinking, calculations, and orientation. It contains the same items as the original MoCA except those requiring visual abilities have been removed as this is administered over the phone. Time to administer the MoCA- BLIND is approximately 5-10 minutes. The total possible score is 22 points; a score of 19 or above is considered normal.
WMS-R: Wechsler Memory Scale-Logical Memory I & II | Change in score from baseline to post-intervention 6 months
  Logical Memory I & II will be used to assess episodic memory. A brief story will be read to the participant who will then asked to retell it immediately (I) and after a 10- min delay filled with other activities (II). The score is the number of the 25 story units recalled immediately (I) and after the delay (II).
Stroop Neuropsychological Screening Test (Trennerry et al., 1989) | Change in score from baseline to post-intervention 6 months
  Stroop Test will be used to assess executive function. In Stroop C, participants are shown a list of colors printed in conflicting color ink and are asked to read words (names of colors). The second part of this task is Stroop CW in which participants are shown a list of colors printed in conflicting color ink and are asked to say the color of the ink the word is printed. The scores are the number of words named correctly in 30 seconds and the number of colors named correctly in 30 seconds subtracting the number of errors. respectively.
Digit Span Test (Wechsler, 1987) | Change in score from baseline to post-intervention 6 months
  Digit Span Forward & Backward will be used to assess working memory. Digit strings of increasing length will be read, and the participant is asked to repeat each string forward (Digit Span Forward) or backward (Digit Span Backward). The score is the number of correctly retrieved strings in each part.
Word fluency Test (Welsh et al., 1994) | Change in score from baseline to post-intervention 6 months
  Word Fluency will be used to assess executive function. The Word Fluency Test asks participants to name as many animals (part 1) or fruits and vegetables (part 2) as possible in 60 seconds. The score is the sum of the number of animals and the number of fruits and vegetables named.
Digit Ordering Test (Cooper at al., 1991) | Change in score from baseline to post-intervention 6 months
  Digit ordering test will be used to assess working memory. For Digit Ordering, digit strings of increasing length will be read and the participant is asked to reorder the digits and say them in ascending order. The score is the number of correctly reordered strings.

SECONDARY OUTCOMES:
Minutes per day of light and moderate-to-vigorous physical activity via GT3x Actigraph Accelerometer | Change in minutes per day of light and moderate-to-vigorous physical activity from baseline to post-intervention 6 months
  Device-assessed physical activity via GT3x Actigraph accelerometers will be used to assess minutes per day spent in light physical activity and moderate-to-vigorous physical activity.
Godin-Shephard leisure-time physical activity questionnaire (GLTEQ) | Change in activity score from baseline to post-intervention 6 months
  The GLTEQ is a 3-item questionnaire that assesses the number of times in the past week an individual participates in strenuous (eg, jogging), moderate (eg, brisk walking), and mild (eg, easy walking) exercise of more than 15 minutes in duration. Frequencies from the strenuous and moderate items are multiplied by 9 and 5 metabolic equivalents, respectively, and summed to calculate a moderate-to-vigorous activity score in accordance with the GLTEQ scoring protocol.
MIND diet adherence | Change in MIND diet adherence from baseline to post-intervention 6 months
  Block 2005 Food Frequency Questionnaire will be used to compute MIND diet scores. Frequency of consumption for food items was assigned a score of 0, 0.5, or 1, where scores ranged from 0 (lowest adherence) to 15 (highest adherence).
National Institutes of Health (NIH) Toolbox: Perceived Stress Fixed Form Age 18+ v2.0 | Change in scores from baseline to post-intervention 6 months
  NIH Tool box measure of perceived stress is a self-reported measure that assesses how unpredictable, uncontrollable, and overloaded respondents find their lives. 10 items are administered using a 5-point scale, with options ranging from "never" to "very often". Higher scores are indicative of higher perceived stress.
National Institutes of Health (NIH) Toolbox General Life Satisfaction Fixed Form A Age 18+ v2.0 | Change in scores from baseline to post-intervention 6 months
  NIH Tool box measure of general life satisfaction assesses global feelings and attitudes about one's life. 5 items are administered using a 5 and 7-point scale, ranging from "strongly disagree" to "strongly agree". Higher scores are indicative of higher general life satisfaction.
National Institutes of Health (NIH) Tool Box: Sadness Fixed Form Age 18+ v2.0 | Change in scores from baseline to post-intervention 6 months
  NIH Toolbox measure of depression/sadness assesses negative mood, negative views of self, and negative social cognition. 8 items are administered using a 5-point scale ranging from "never" to "always". Higher scores are indicative of more sadness.
National Institues of Health (NIH) Toolbox Loneliness Fixed Form Age 18+ v2.0 | Change in scores from baseline to post-intervention 6 months
  NIH Toolbox measure of loneliness assesses perceptions of loneliness using 5 items, responses from a 5-point scale ranging from "never" to "always". Higher scores are indicative of more loneliness.
Spectroscopy-Based Veggie Meter® | Change in scores from baseline to post-intervention 6 months
  The Veggie Meter (VM; Longevity Link Inc., Salt Lake City, UT, USA) is a commercially available device that uses reflection spectroscopy to measure the level of carotenoid pigments in a person's skin by scanning the tip of the finger. Scores range from 0-800.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Hughes, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Urbana-Champaign, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: No